CLINICAL TRIAL: NCT03336957
Title: Effect of Non-Surgical Periodontal Therapy on Pregnancy-Related Degree of Gingival Inflammation and Stress Markers
Brief Title: Stress and Gingival Inflammation in Non-pregnant and Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Ozge Gokturk, Principal Investigator, Tokat Gaziosmanpasa University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-KAEK-154
Record Dates: First submitted 2017-11-02; First posted 2017-11-08 (Actual); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Periodontal Diseases; Pregnancy Gingivitis
Keywords: chromogranin A, stress, gingivitis, pregnancy
MeSH Terms: conditions — Periodontal Diseases; Gingivitis | interventions — Periodontal Index

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant group (Experimental): Test group, non-surgical periodontal therapy (NPT) consisted of scaling and oral hygiene instruction was applied. IL- 1β AND IL-10 in the GCF and Cg A in saliva samples were taken before and after periodontal treatment.
  Interventions: Procedure: periodontal treatment
- Non-Pregnant (Active Comparator): Control group, non-surgical periodontal therapy (NPT) consisted of scaling and oral hygiene instruction was applied. IL- 1β AND IL-10 in the GCF and Cg A in saliva samples were taken before and after periodontal treatment.
  Interventions: Procedure: periodontal treatment

INTERVENTIONS:
Procedure: periodontal treatment — non-surgical periodontal therapy (NPT) consisted of scaling, root planning, and oral hygiene instruction

SUMMARY:
Background: The purpose of the present study is to research whether stress scale scores alter with relationship to gingival inflammation and examine the impact of non-surgical periodontal therapy during pregnancy on the levels of cytokines in gingival crevicular fluid (GCF) and on salivary stress-related hormones.

Methods: 30 non-pregnant (control group) and 30 pregnant women (test group) who fulfilled the study inclusion criteria were chosen. The participants with moderate/severe gingivitis were included. Clinical data and samples of GCF and salivary were collected at baseline and after periodontal therapy. The levels of cytokines interleukin-1 beta (IL-1β) and IL-10, and concentration of salivary chromogranin A (Cg A) hormone were analyzed by enzyme-linked immunosorbent assay kits.

DETAILED DESCRIPTION:
Periodontal clinical measurements and periodontal treatment were applied by a previously trained and calibrated examiner. Clinical parameters measurements including; probing pocket depths (PPD; the distance from the gingival margin to the base of the gingival sulcus), clinical attachment level (CAL), full mouth gingival index (GI)21 and plaque index (PI)20 scores using a periodontal probe were registered following saliva and GCF sample collection. Then, non-surgical periodontal therapy (NPT) consisted of scaling, root planning, and oral hygiene instruction was applied. Clinical measurements, recruitment of GCF, and saliva samples were repeated after three weeks.

Gingival Crevicular Fluid and Saliva Sample Collection Selected anterior teeth for GCF sampling were isolated from saliva using cotton rolls, a gentle stream of air was conducted parallel to the root surface for 5 to 10 seconds to dry the area.

The periopaper strips were gently inserted into the gingival crevice until resistance was felt and were left in place for 30 s and were collected from mesio-buccal sulcus of teeth in the anterior region of each patient (two samples per patient and per visit). The samples containing blood were discarded and were placed in sterile Eppendorf tubes and were stored at -20°C until the assay procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Must be systemically healthy;
2. Must be at least twenty teeth in the mouth;
3. Clinical diagnosis of gingivitis;
4. Must be the probing pocket depth (PPD)≤3 mm in all four quadrants.

Exclusion Criteria:

* the use of anti-inflammatory,
* antimicrobial and hormone therapy within the preceding 6 months,
* having psychiatric disorders,
* a systemic disease,
* smoking cigarettes and
* for the control group breastfeeding, pregnancy and menstrual periods.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2016-06-01; Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
salivary Cg A hormone concentration | up to 8 weeks
  Samples should be taken before and after treatment and evaluated using ELISA kits

SECONDARY OUTCOMES:
IL-1β and IL-10 Cytokine levels in the GCF | up to 8 weeks
  Samples should be taken before and after treatment and evaluated using ELISA kits

IPD SHARING:
Plan to Share IPD: Undecided
individual participant data for all primary and secondary outcome measures will be made available.

REFERENCES:
- [Derived] Yarkac FU, Gokturk O, Demir O. Effect of non-surgical periodontal therapy on the degree of gingival inflammation and stress markers related to pregnancy. J Appl Oral Sci. 2018 Jul 23;26:e20170630. doi: 10.1590/1678-7757-2017-0630. PMID 30043934